CLINICAL TRIAL: NCT02095964
Title: HDL-Cholesterol is Inversely Related With Inflammation in Cardiac Syndrome X
Brief Title: HDL-C in Cardiac Syndrome X
Acronym: HIRICS-X
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BYIEAH-281
Record Dates: First submitted 2014-03-17; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Ischaemia; Unstable Angina; Microvascular Angina
Keywords: cardiac syndrome X; inflammation; dyslipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease; Angina, Unstable; Microvascular Angina; Inflammation; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cardiac Syndrome X
- Control Group

SUMMARY:
High density lipoprotein cholesterol (HDL-C) is in the centrum of the process of reverse cholesterol transport from peripheral cells to the liver[10]. HDL-C promotes endothelial generation of nitric oxide (NO) and improves endothelial function and arterial vasoreactivity[11]. In several studies, lower HDL-C level was reported to be associated with increased coronary artery disease (CAD) risk[12-14]. HDL-C also has anti- inflammatory and anti-oxidant activities[15,16]. Concerning anti-inflammatory activity, HDL-C inhibits the activation of monocytes/macrophages and neutrophils[17,18] and inhibits the expression of endothelial adhesion molecules, such as vascular cell adhesion molecule-1 (VCAM-1) and E-selectin[15].

In this study we aimed to investigate the relation of HDL-C level with systemic inflammatory markers in patients with cardiac syndrome X (CSX).

ELIGIBILITY:
Inclusion Criteria:

* Must be able to get exercise stress test
* Must be able to have coronary angiography
* Clinical diagnosis of typical anginaduring rest or effort
* Abnormal test result for exercise ECG or myocardial perfusion scintigraphy
* Must have of angiographically normal epicardial coronary arteries

Exclusion Criteria:

* Patients with valvular heart disease (mitral stenosis and moderate to severe mitral regurgitation
* Patients with moderate to severe aortic stenosis and regurgitation including mitral annular calcification)
* Patients with heart failure (left ventricular ejection fraction <50%)
* Patients with congenital heart disease, cardiomyopathy, left ventricular hypertrophy, right ventricular hypertrophy
* Patients with cardiac surgery
* Patients with thyroid disease
* Patients with anemia
* Patients with pulmonary diseases
* Patients with infectious diseases (locally or systemic)

Ages: 47 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: CSX was defined as typical chest pain during rest or effort, abnormal test result for exercise ECG and myocardial perfusion scintigraphy, and the presence of angiographically normal epicardial coronary arteries. Control group was selected from volunteers presented to our hospital with the complaint of typical anginal chest pain who had no ischemia on myocardial perfusion scintigraphy or during the treadmill exercise test, had similar risk profile with the patients (diabetes, hypertension, age, gender) and had normal epicardial coronaries at coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
HDL-Cholesterol | 6 MONTHS
  HDL-Cholesterol <40 mg/dL(male) / < 50mg/dL(female) ==> low HDL-C
Cardiac Syndrome X | 6 months
  Patients who have typical anginal chest pain+ischaemic findings at exercise stress test/myocardial scintigraphy + normal epicardial coronaries at coronary angiography ==> Cardiac syndrome X
Inflammation | 6 months
  CRP > 2,98 mg/dL ==> systemic inflammation